CLINICAL TRIAL: NCT05499936
Title: Peking Union Medical College Hospital
Brief Title: 68Ga-FAPI PET/CT for the Detection of Adenoid Cystic Carcinoma(ACC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHFAPI-ACC
Record Dates: First submitted 2022-06-28; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2021-10

CONDITIONS: 68Ga-FAPI PET/CT; Metastatic Adenoid Cystic Carcinoma
Keywords: 68Ga-FAPI; PET/CT; Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI PET/CT (Experimental): Imaging was performed 30-60 minutes after injection of 2-4mci 68Ga-FAPI tracer
  Interventions: Drug: 68Ga-FAPI

INTERVENTIONS:
Drug: 68Ga-FAPI — 68Ga-FAPI were injected into the patients before the PET/CT scans

SUMMARY:
This study was used to study the diagnostic value of 68Ga-FAPI, a novel fibroblast activating inhibitor, in metastatic adenoid cystic carcinoma（ACC）

DETAILED DESCRIPTION:
68Ga-FAPI is a positron labeled inhibitor of fibroblast activating protein, which has been widely used in malignant tumor imaging in recent years. Adenoid cystic carcinoma (ACC) is a rare epithelial malignant tumor, which usually originates from salivary glands. Its typical characteristics are long clinical course and high rate of distant metastasis. The purpose of this study was to investigate the clinical value of 68Ga Fapi pet/ct in metastatic adenoid cystic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* patients with ACC suspected metastatic tumor,and being able to provide basic information and sign the written informed consent form

Exclusion Criteria:

* claustrophobia, pregnancy, breastfeeding, kidney or liver failure, inability to fulfill the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-FAPI in ACC | 1 year
  The maximum and mean standard uptake values (SUVmax and SUVmean) were measured in the background of lesion, liver, muscle and mediastinal blood pool, respectively.

SECONDARY OUTCOMES:
lesions detected by 68Ga-FAPI PET/CT | 1 year
  The number of target lesions in each organ system was calculated by 68Ga-FAPI PET/CT

OTHER OUTCOMES:
compared with 18F-FDG PET/CT or other imaging like CT and MRI | 1 year
  The number of lesions detected by 68Ga-FAPI PET/CT was compared with 18F-FDG PET/CT or other imaging like CT and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, China